CLINICAL TRIAL: NCT04428073
Title: A Phase I Trial of a Therapeutic Vaccine (Covax-19™) in SARS-CoV-2 Infected Patients
Brief Title: Therapeutic Vaccine Trial of COVID-19 for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GeneCure Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GC004
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: COVID
Keywords: SARS-CoV-2; COVID-19; therapeutic vaccine
MeSH Terms: conditions — COVID-19 | interventions — SARS-CoV-2 recombinant spike protein with delta inulin and CpG-ODN adjuvant vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose group (Experimental): Subjects will receive 1.0 mL of low dose vaccine at week 0 and 2.
  Interventions: Biological: Covax-19™
- High dose group (Experimental): Subjects will receive 1.0 mL of high dose vaccine at week 0 and 2.
  Interventions: Biological: Covax-19™

INTERVENTIONS:
Biological: Covax-19™ — Therapeutic vaccine for SARS-CoV-2 infection

SUMMARY:
GC004 is a Phase I trial to evaluate the safety and the immune responses of a therapeutic vaccine in SARS-CoV-2 infected patients. Covid-19 confirmed patients with mild or no symptoms will be enrolled sequentially into low dose and high dose groups. Following the vaccination subjects who received at least one vaccination will be followed for safety through week 26.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of Covid-19 infection based on laboratory evidence of positivity by RT- PCR.
2. Patients who have no clinical symptoms (fever, cough and dyspnea).
3. Patients who have mild clinical symptoms that could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath (dyspnea).
4. Screening laboratory values within institutional normal range or judged to be not clinically significant by clinical investigator.
5. Ability and willingness of subject to give written informed consent.
6. Negative pregnancy test on the day prior to each vaccination.
7. Willingness to use adequate contraception by study participants.

Exclusion Criteria:

1. History of respiratory and cardiovascular diseases, hematologic disease (e.g., cryoglobulinemia, lymphoma), renal disease, dermatologic disease (e.g., lichen planus, porphyria cutanea tarda).
2. Autoimmune diseases or clinically serious cardiac, pulmonary, gastrointestinal, hepatic, renal or neurologic disease, which in the opinion of the investigator will compromise ability to participate in the study.
3. Pregnancy and breast-feeding.
4. Prior or current systemic cancer chemotherapy.
5. Investigational agents and immunomodulators (cyclosporine, hematological growth factors, systemic corticosteroids, interleukins or interferons) within 90 days prior to study entry.
6. Anaphylaxis or allergy to vaccine components.
7. Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
8. Any other serious diseases other than Covid-19 infection including current or recent (within 5 years) cancers.
9. Subjects who are immunocompromised or immunosuppressed due to disease or medications.
10. Women who are lactating.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of a therapeutic Covid-19 vaccine in participants by measuring the severity of local and systemic adverse events and laboratory abnormalities. | 26 weeks
  Frequency and severity of adverse events, laboratory abnormalities, local and systemic reactogenicity, signs and symptoms after vaccinations.

SECONDARY OUTCOMES:
To evaluate the immunogenicity of a therapeutic Covid-19 vaccine in participants by measuring CD8+ T cells immune response | 6 weeks
  Magnitude of IFN-γ producing CD8+ T cells to SARS-CoV-2 nucleocapsid peptides pools after vaccinations.
Virologic response after vaccination | 4 weeks
  Detection of SARS-CoV-2 by RT-PCR in respiratory tract specimens at week 0, 1, 2, 3, and 4.
Clinical outcome and progression after vaccinations | 6 weeks
  Number of participants with moderate, severe or critical Covid-19 at week 6.

IPD SHARING:
Plan to Share IPD: No
The final study results will be published in peer reviewed journals.